CLINICAL TRIAL: NCT06617273
Title: Near Normal Intraocular Pressure Cataract Surgery in Patients with Diabetic Retinopathy Using Active Anterior Chamber Pressure Sensing and Regulation - a Randomized Controlled Comparative Clinical Trial
Brief Title: Cataract Surgery with Near Normal Eye Pressure in Patients with Diabetic Retinopathy
Acronym: NNIOP-PHACO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNIOP-PHACO
Record Dates: First submitted 2024-09-11; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Retinopathy; Cataract
Keywords: Diabetic Retinopathy; Phacoemulsification; Microincision Phacoemulsification; Cataract; Intraocular pressure; Active anterior chamber pressure
MeSH Terms: conditions — Diabetic Retinopathy; Cataract

STUDY DESIGN:
Intervention Model Description: controlled randomized, comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A) IOP 28mmHg on the better eye and IOP 50mmHg on the worse eye (Other): Near normal intraocular pressure cataract surgery using active anterior chamber pressure sensing and regulation
  Interventions: Device: Ophthalmosurgical handpiece with active anterior chamber pressure sensing and regulation
- B) IOP 28mmHg on worse eye and IOP 50mmHg on the better eye (Other): Near normal intraocular pressure cataract surgery using active anterior chamber pressure sensing and regulation
  Interventions: Device: Ophthalmosurgical handpiece with active anterior chamber pressure sensing and regulation

INTERVENTIONS:
Device: Ophthalmosurgical handpiece with active anterior chamber pressure sensing and regulation — Cataract surgery in patients with diabetic retinopathy using active anterior chamber pressure sensing and regulation

SUMMARY:
Diabetes mellitus is a chronic metabolic disease that can lead to visual impairment and eye complications such as diabetic retinopathy and diabetic macular edema. Diabetics are considered a vulnerable patient group for cataract surgery, as microincision phacoemulsification (MICS) in diabetics is associated with a higher risk of postoperative swelling of the macula and cornea (macular or corneal edema). In addition, the ultrasound energy emitted during MICS, high and fluctuating intraocular pressure and the movement of surgical instruments and lens material are the main causes of surgical trauma. The medical device "Centurion Vision System" with the "Active Sentry" handpiece was developed specifically to improve the stability of the anterior chamber during surgery and to enable operations at low, almost normal physiological intraocular pressure settings.

The central question of the study is therefore, whether a stable intraocular pressure close to physiological normal conditions (28 mmHg) during surgery can lead to a reduction in surgical trauma. In this prospective and randomized study, patients suffering from diabetes and having a planned bilateral MICS are included in one of two study arms:

A) The participant is operated on with an IOP of 28 mm Hg in the better eye and an IOP of 50 mm Hg in the worse eye or B) the participant is operated on with an IOP of 28 mm Hg in the worse eye and an IOP of 50 mm Hg in the better eye.

ELIGIBILITY:
Inclusion Criteria:

1. Indication for immediate sequential bilateral microincision cataract surgery
2. Diagnosis of Diabetes Mellitus treated with oral medication or insulin therapy and confirmed by HbA1c ≥6,5 %
3. Presence of diabetic retinopathy grade ≥1 on the international clinical diabetic retinopathy (ICDR) severity scale
4. LOCS 2-4 with no more than 1 grade difference between both eyes
5. Male or female patient aged 50 - 85 years of age at time of consent
6. Understands and agrees to comply with the study procedures and provides written informed consent as documented by signature

Exclusion Criteria:

1. Participation in another clinical trial within 30 days before pre-screening and throughout the trial
2. Prior intraocular surgery of any type
3. History of diabetic macular edema
4. Presence of macular edema, defined as central retinal thickness of >300 µm plus intraretinal or subretinal fluid on OCT within range of 1mm of foveal center
5. Presence of any retinal or choroidal disease, other than diabetes, that could affect retinal thickness
6. Known history of uveitis
7. Documented use of systemic or topical steroid or other immunosuppressive medication within the last 3 months
8. ACF >10 ph/ms. ACF difference between right and left eye > 4ph/ms
9. Difference of DRP grading between right and left eye of more than 1 grade (ICDR)
10. Inability to measure total macular volume due to, but not limed to, too dense cataract, vitreous bleeding
11. Woman of childbearing potential (WOCBP) who is breastfeeding, has a positive urine pregnancy test, is not willing to undergo a urine pregnancy test upon entering or exiting the study, intends to become pregnant during the study, or does not agree to use adequate birth control methods for the duration of the study
12. Patients in possession of an active implantable medical device (AIMD)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Delta ACF | 1 week
  Difference from pre- to postoperative ACF (delta ACF) at day 1 (FU1) and day 7 (FU2) after cataract surgery.

SECONDARY OUTCOMES:
BCVA | 1 month
  Difference between pre- to postoperative BCVA
5mm corneal volume | 1 month
  Pentacam derived
Anterior chamber depth | 1 month
  Pentacam derived
Mydriatic pupil width | 1 month
  Pentacam derived
Endothelial cell density | 1 month
  Quantifying assessment of endothelial cell loss via specular microscopy; (28 +-3) days after surgery.
Assessment of intraoperative complications | 1 month
  Screening for the presence of posterior capsular ruptures
Assessment of postoperative complications | 1 month
  Presence of cystoid macular edema
Intraoperative events | Day 0 (Surgery)
  Assessment of any event in regard to phacoemulsification settings
Central macular thickness | 1 month
  Pre- and postoperative assessment of central macular thickness via optical coherence tomography (OCT)
Total macular volume | 1 month
  Pre- and postoperative assessment of total macular volume via optical coherence tomography (OCT)
Retinal Nerver fiber layer thickness (RNFL) | 1 month
  Pre- and postoperative assessment of RNFL via optical coherence tomography (OCT)
Central corneal thickness | 1 month
  Pre- and postoperative assessment of central corneal thickness via optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, University Hospital for Ophthalmology and Optometry, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No